CLINICAL TRIAL: NCT04565340
Title: Foley Catheter Versus Prostaglandin E2 (Propess) Inserts for Induction of Labor in Women With Term Premature Rupture Of Membranes : Mode of Delivery and Maternal and Fetal Outcomes
Brief Title: Foley vs Propess for Induction of Labor in Women With Term PROM : Mode of Delivery, Maternal and Fetal Outcomes
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0143
Record Dates: First submitted 2020-09-14; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Premature Rupture of Membranes at Term; Mode of Delivery
Keywords: Complications and outcomes maternal and neonatal; Induction of labor; Prostaglandins; Foley Catheter
MeSH Terms: interventions — Parturition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Induction of labor with Foley catheter: Induction of labor with Foley catheter
- Induction of labor with Propess: Induction of labor with Propess
  Interventions: Other: Mode of delivery, maternal and neonatal outcomes/complications

INTERVENTIONS:
Other: Mode of delivery, maternal and neonatal outcomes/complications — Mode of delivery, maternal and neonatal outcomes/complications
  Groups: Induction of labor with Propess

SUMMARY:
Premature rupture of membranes at term is a rupture that occurs at term (>37SA) before the start of labor. It complicates 5 to 10% of pregnancies and 6 to 22% of term pregnancies.

Althought some studies support efficacy of the Foley catheter for cervical ripening at term in induction of labor with intact membranes, it has not been well studied in women with premature rupture of membranes at term.

The aim of this retrospective study at the Montpellier University Hospital is to evaluate the effect of the Foley catheter compared to Propess in women with premature rupture of membranes at term, on the induction of labor and the maternal and fetal complications.

ELIGIBILITY:
Inclusion criteria:

* Singleton Pregnancy >37 weeks of gestation
* Premature Rupture Of Membranes
* Cephalic presentation
* Unfavorable cervix (BISHOP <7)
* No contraindication of induction methods

Exclusion criteria:

* Multiple gestation
* PROM with spontaneous labor
* Induction of labor with both methods
* Previous cesarean section
* Unexplained metrorrhagia / Placenta praaevia
* Suspected intraamniotic infection
* Herpes simplex virus
* Human immunodeficiency virus
* Any contraindication to vaginal delivery
* Latex allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with Premature Rupture Of Membranes at term (>37SA) at Montpellier University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
mode of delivery (vaginal delivery or cesarean) | 1 day
  mode of delivery (vaginal delivery or cesarean)

SECONDARY OUTCOMES:
maternal and fetal outcomes | 1 day
  looking for maternal complications (endometritis, chorioamniotitis, transfusion, post-partum hemorrhage) and neonatal complications (sepsis, apgar<7 at 5minutes, pH <7,15, neonatal intensive care unit)

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PUPH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC